CLINICAL TRIAL: NCT01848002
Title: A Randomized, Placebo-Controlled, Double-Blind, Multi-dose Study of the Safety and Pharmacokinetics of Recombinant Factor XIII Administration in Healthy Volunteers
Brief Title: Safety and Pharmacokinetics of Recombinant Factor XIII Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F13-1662
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Congenital Bleeding Disorder; Congenital FXIII Deficiency; Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rFXIII (Experimental)
  Interventions: Drug: catridecacog
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: catridecacog — For 5 consecutive days, one daily dose of rFXIII was administered intravenously (IV) to eight subjects in each dose group (10 or 25 U/kg).
  Arms: rFXIII
Drug: placebo — For 5 consecutive days, one daily dose of placebo was administered intravenously (IV) to two subjects in each dose group (10 or 25 U/kg).
  Arms: Placebo

SUMMARY:
This trial was conducted in Europe. The aim of this trial was to investigate safety and pharmacokinetics of multiple doses of catridecacog (recombinant factor XIII, rFXIII) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Normal platelet count and clotting parameters
* Adequate renal and hepatic function
* Negative serum pregnancy test within 21 days prior to enrollment and negative urine pregnancy test on admission to the clinical research unit (if subject female and of child-bearing potential)
* Agreement to use a medically accepted form of contraception from the time of enrollment to completion of all follow-up study visits (if subject a sexually active male or female of childbearing potential)
* Negative drug and negative alcohol screens

Exclusion Criteria:

* Known antibodies or hypersensitivity to FXIII
* Known bleeding or hematologic disorder
* Known allergy to yeast
* Receipt of blood products within 30 days of screening
* Donation of blood within 30 days prior to enrollment
* Surgical procedure of any type within 30 days prior to enrollment
* History of autoimmune disorders involving autoantibodies, e.g., systemic lupus erythematosus
* Treatment with any experimental agent within 30 days of study enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-05; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Days 0-33

SECONDARY OUTCOMES:
Incidence of clinically significant changes from baseline in physical examination or laboratory measurements | From days -1 through day 33
Incidence of rFXIII antibodies, as measured by ELISA (Enzyme-Linked Immuno Sorbent Assay) | From days -1 through day 33
Incidence of yeast antibodies | From days -1 through day 33

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Berkshire, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com